CLINICAL TRIAL: NCT02649946
Title: A Prospective, Multi-Center, Randomized, Concurrently-Controlled Clinical Study of the BARD® COVERA™ Arteriovenous (AV) Stent Graft in the Treatment of Stenosis in the Venous Outflow of AV Fistula Access Circuits (AVeNEW)
Brief Title: Clinical Study of the BARD® COVERA™ Arteriovenous (AV) Stent Graft
Acronym: AVeNEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPV-14-005
Record Dates: First submitted 2016-01-04; First posted 2016-01-08 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Stenosis; Restenosis
Keywords: ESRD; Stenosis; Restenosis; Hemodialysis; AV Fistula; Arteriovenous (AV)
MeSH Terms: conditions — Constriction, Pathologic; Kidney Failure, Chronic; Arteriovenous Fistula | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Covera Vascular Covered Stent following PTA (Experimental): Placement of the Covera Vascular Covered Stent following percutaneous transluminal angioplasty (PTA)
  Interventions: Device: Covera Vascular Covered Stent following PTA
- PTA only using uncoated PTA Balloon (Active Comparator): Percutaneous Transluminal Angioplasty (PTA) will be performed using a commercially available uncoated PTA balloon. Balloons with an external wire support, cutting/scoring component or other similar modifications are not permitted. Multiple balloons, inflations and/or prolonged inflation may be used.
  Interventions: Procedure: Percutaneous Transluminal Angioplasty (PTA) with Uncoated PTA Balloon

INTERVENTIONS:
Device: Covera Vascular Covered Stent following PTA — Treatment of stenoses with primary percutaneous transluminal angioplasty (PTA) and placement of the Covera Vascular Covered Stent.
  Arms: Covera Vascular Covered Stent following PTA
Procedure: Percutaneous Transluminal Angioplasty (PTA) with Uncoated PTA Balloon — Treatment of stenoses with PTA only
  Other Names: Standard Balloon Angioplasty (POBA)
  Arms: PTA only using uncoated PTA Balloon

SUMMARY:
The objective of this study is to assess the safety and effectiveness of the COVERA™ Vascular Covered Stent for the treatment of stenotic lesions in the upper extremity venous outflow of the Arteriovenous (AV) access circuit.

DETAILED DESCRIPTION:
This study will compare the use of the COVERA™ Vascular Covered Stent (following percutaneous transluminal angioplasty (PTA)) to PTA alone for the treatment of stenotic lesions in the upper extremity venous outflow of the arteriovenous (AV) access circuit of subjects dialyzing with an AV fistula.

ELIGIBILITY:
Clinical Inclusion Criteria:

* Subject must voluntarily sign and date the Informed Consent Form (ICF) prior to collection of study data or performance of study procedures.
* Subject must be either a male or non-pregnant female ≥ 21 years of age with an expected lifespan sufficient to allow for completion of all study procedures.
* Subject must be willing to comply with the protocol requirements, including the clinical and telephone follow-up.
* Subject must have an upper extremity arteriovenous (AV) fistula that has undergone at least one successful dialysis session with two-needle cannulation, prior to the index procedure.

Angiographic Inclusion Criteria:

* Subject must have angiographic evidence of a stenosis ≥ 50% (by visual estimation) located in the venous outflow of the AV access circuit and present with clinical or hemodynamic evidence of AV fistula dysfunction.
* The target lesion must be ≤ 9cm in length. Note: multiple stenoses may exist within the target lesion.
* The reference vessel diameter of the adjacent non-stenotic vein must be between 5.0 and 9.0mm.

Clinical Exclusion Criteria:

* The subject is dialyzing with an AV graft.
* The target lesion has had a corresponding thrombosis treated within 7 days prior to the index procedure.
* The hemodialysis access is located in the lower extremity.
* The subject has an infected AV fistula or uncontrolled systemic infection.
* The subject has a known uncontrolled blood coagulation/bleeding disorder.
* The subject has a known allergy or hypersensitivity to contrast media which cannot be adequately pre-medicated.
* The subject has a known hypersensitivity to nickel-titanium (Nitinol) or tantalum.
* The subject has another medical condition, which, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.
* The subject is currently participating in an investigational drug or another device study that has not completed the study treatment or that clinically interferes with the study endpoints. Note: Studies requiring extended follow-up visits for products that were investigational, but have since become commercially available, are not considered investigational studies.

Angiographic Exclusion Criteria:

* Additional stenotic lesions (≥ 50%) in the venous outflow that are > 3cm from the edge of the target lesion and are not successfully treated (defined as < 30% residual stenosis) prior to treating the target lesion.
* An aneurysm or pseudoaneurysm is present within the target lesion.
* The location of the target lesion would require the COVERA™ Vascular Covered Stent be deployed across the elbow joint.
* The target lesion is located within a stent.
* The location of the target lesion would require that the COVERA™ Vascular Covered Stent be deployed at or across the segment of fistula utilized for dialysis needle puncture (i.e., "cannulation zone").
* The location of the target lesion would require that the COVERA™ Vascular Covered Stent be placed in the central veins (subclavian, brachiocephalic, superior vena cava (SVC)) or under the clavicle at the thoracic outlet.
* There is incomplete expansion of an appropriately sized angioplasty balloon to its expected profile, in the operator's judgment, during primary angioplasty at the target lesion prior to randomization.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Dolmatch, M.D., Principal Investigator — The Palo Alto Medical Foundation
Locations (24):
- United States (16):
  - Southwest Vascular Center, Tempe, Arizona
  - Alliance Research Centers, Laguna Hills, California
  - Radiology Imaging Associates, Englewood, Colorado
  - Yale University & Yale New Haven Hospital, New Haven, Connecticut
  - Nephrology Associates, P.A., Newark, Delaware
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Ocala Kidney Group, Ocala, Florida
  - Chicago Access Care, Chicago, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Renal and Transplant Associates of New England, P.C., West Springfield, Massachusetts
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - NC Nephrology, Raleigh, North Carolina
  - Providence Access Care, Providence, Rhode Island
  - Tarrant Vascular Clinic, Fort Worth, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
- Australia (2):
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Adelaide Hospital, Kensington Gardens, South Australia
- LKH-Univ. Klinikum Graz, Graz, Austria
- University Hospital Leuven, Leuven, Vlaams-Brabant, Belgium
- Universitätsklinikum Würzburg, Würzburg, Germany
- Maastricht Universitair Medish Centrum, Maastricht, Netherlands
- Middlemore Hospital, Auckland, New Zealand
- Universitaets Spital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Dolmatch B, Cabrera T, Pergola P, Balamuthusamy S, Makris A, Cooper R, Moore E, Licht J, Macaulay E, Maleux G, Pfammatter T, Settlage R, Cristea E, Lansky A; AVeNEW Trial Investigators. Prospective, randomized, multicenter clinical study comparing a self-expanding covered stent to percutaneous transluminal angioplasty for treatment of upper extremity hemodialysis arteriovenous fistula stenosis. Kidney Int. 2023 Jul;104(1):189-200. doi: 10.1016/j.kint.2023.03.015. Epub 2023 Mar 27. PMID 36990214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 9, 2016, and July 20, 2017, Investigators randomized 280 subjects into the study at 24 sites in the US, Europe, and Australia/New Zealand (50-75% of subjects treated in the US). The final subject completed 6 month follow-up on January 30, 2018. Anticipated data of study completion (last subject, last visit) is Q3, 2019.
Period: Overall Study
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Started | 142 | 138
Completed | 130 | 123
Not Completed | 12 | 15
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 7 | 9
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Erroneously enrolled | 1 | 0
Not completed — Missed 6-month follow-up visit | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon | Total
Number analyzed (Participants) | 142 | 138 | 280
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 79 | 76 | 155
  ≥ 65 and < 75 years | 36 | 45 | 81
  ≥ 75 years | 27 | 17 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 107
  Male | 89 | 84 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 54 | 102
  Not Hispanic or Latino | 93 | 84 | 177
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 6 | 6
  Black or African American | 36 | 36 | 72
  Native Hawaiian or Other Pacific Island | 2 | 0 | 2
  White | 100 | 92 | 192
  Other | 4 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants] — Please note that New Zealand sites are included in the Australia section.
  Participants
    United States | 131 | 131 | 262
    Europe | 7 | 3 | 10
    Australia | 4 | 4 | 8
Medical History [Count of Participants; unit: Participants] — Medical history information, including medical risk factors as well as selected medical history background for the ITT population is provided. "Other Disease" category includes Bleeding Disorder, Cancer, Steal Syndrome, and other.
  Participants
    Diabetes (Type 1 and 2) | 108 | 103 | 211
    Dyslipidemia | 95 | 85 | 180
    Hypertension | 139 | 133 | 272
    Cigarette Smoking (current or former) | 62 | 62 | 124
    Cardiovascular Disease | 95 | 95 | 190
    Other Disease | 129 | 129 | 258
AV Access Circuit Description: Target Limb [Count of Participants; unit: Participants]
  Left Arm | 106 | 110 | 216
  Right Arm | 36 | 28 | 64
AV Access Circuit Description: Access Position [Count of Participants; unit: Participants]
  Forearm | 9 | 8 | 17
  Upper Arm | 132 | 130 | 262
  At Elbow | 1 | 0 | 1
AV Access Circuit Description:Inflow Artery [Count of Participants; unit: Participants]
  Axillary | 2 | 2 | 4
  Brachial | 128 | 127 | 255
  Radial | 12 | 9 | 21
AV Access Circuit Description: Outflow Vein [Count of Participants; unit: Participants]
  Axillary | 2 | 1 | 3
  Basilic | 35 | 42 | 77
  Cephalic | 105 | 95 | 200
AV Access Circuit Description: Fistula Configuration [Count of Participants; unit: Participants]
  Radiocephalic | 12 | 9 | 21
  Brachiocephalic | 84 | 78 | 162
  Transposed Brachiobasilic | 27 | 37 | 64
  All Other | 19 | 14 | 33
AV Access Circuit Description: Transposed [Count of Participants; unit: Participants]
  Yes | 36 | 43 | 79
  No | 106 | 95 | 201

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness Endpoint: Number of Participants With Target Lesion Primary Patency (TLPP)
Description: TLPP is defined as the interval following the index intervention until the next clinically driven reintervention at, or adjacent to,the original treatment site or until the extremity is abandoned for permanent access. Primary patency ends when any of the following occurs: a) clinically driven reintervention in the treatment area; b) thrombotic occlusion within the treatment area; c) surgical intervention that excludes the original treatment area from the AV circuit, and/or d) abandonment of the AV fistula due to inability to treat the original treatment area. COVERA Vascular Covered Stent (following PTA) is evaluated against subjects treated PTA alone.
Time Frame: 6 months post index procedure
Population: Number of Participants with Target Lesion Primary Patency. Modified Intended to Treat (mITT) population results were analyzed for this effectiveness endpoint. N = number of subjects in mITT population with evaluable data. Excluded subjects that discontinued, expired and or access abandoned prior to day 15.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 134 | 117
Participants | 105 | 55
Statistical Analysis 1: Comparison: PTA Only Using Uncoated PTA Balloon; Hypothesis: The (survival) rate in subjects treated with the COVERA Vascular Covered Stent (following PTA) with respect to TLPP through 6 months is greater than that in subjects treated with PTA alone in the treatment of stenoses in the upper extremity venous outflow of subjects dializing with an AV fistula. Sample size calculation: 238 randomized subjects [214 evaluable] will give 92% power with one-sided type 1 error = 0.025; Test type: Superiority — TLPP evaluated at 6 months post-index procedure to assess if TLPP of COVERA is superior to that of PTA alone, by direct comparison; p < 0.001, Chi-squared — Test successful if the one-side p-value is less than 0.025 and the result is in favor of the COVERA Vascular Covered Stent

2. Primary Outcome: Number of Participants With Freedom From AV Access Circuit Localized or Systemic Serious Adverse Events
Description: Safety is defined as freedom from any adverse event(s) (AEs), localized or systemic, that reasonably suggests the involvement of the AV access circuit (not including stenosis or thrombosis) that require or result in any of the following alone or in combination: additional interventions (including surgery); in-patient hospitalization or prolongation of an existing hospitalization; or death.
Time Frame: 30 days post index procedure
Population: Number of Participants Free from Primary Safety Events. All Intended to Treat Subjects (ITT) are included in this analysis. Primary safety endpoint evaluated against standard PTA alone.2 subjects excluded from N COVERA due to discontinuation or death prior to day 23 of follow up. One subject excluded from N PTA arm due to death prior to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 140 | 137
Participants | 133 | 132
Statistical Analysis 1: Comparison: PTA Only Using Uncoated PTA Balloon; Hypothesis: The safety rate in subjects treated with the COVERA Vascular Covered Stent (following PTA) is non-inferior to the safety rate in subjects treated with PTA alone through 30 days in the treatment of stenotic lesions. Sample size: 238 randomized subjects [226 evaluable] will give 85% power with one-sided type 1 error = 0.025; Test type: Non-Inferiority — Non-inferiority Farrington and Manning Exact Test is used to test the primary safety hypothesis. The test is successful if the one-sided p-value is less than 0.025; p = 0.0022, Farrington and Manning; Non-inferiority test with non-inferiority margin of 10%

3. Secondary Outcome: Number of Patients With Target Lesion Primary Patency (TLPP) at 12 Months Post Index Procedure
Description: TLPP is defined as the interval following the index intervention until the next clinically driven reintervention at the original treatment site or until the extremity is abandoned for permanent access. Primary patency ends when any of the following occurs: a) clinically driven reintervention in the treatment area; b) thrombotic occlusion within the treatment area; c) surgical intervention that excludes the original treatment area from the AV circuit, and/or d) abandonment of the AV fistula due to inability to treat the original treatment area.
Time Frame: 12 months post-index procedure
Population: Number of Participants with Target Lesion Primary Patency (TLPP). Number of participants (n) in each follow-up periods varies from overall enrollment (N) as some subjects discontinued participation before the 12 month follow-up or did not meet endpoint inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 124 | 114
Participants | 67 | 23

4. Secondary Outcome: Number of Participants With Access Circuit Primary Patency (ACPP).
Description: ACPP is defined as the interval following the index intervention until the next access thrombosis or repeated intervention.
  ACPP ends with a reintervention anywhere within the access circuit. Vessel rupture caused by PTA is not an ACPP failure unless achieving hemostasis also causes thrombosis.
  Testing of this secondary endpoint is performed in a hierarchical fashion. Thus, In order to perform hypothesis test of ACPP at 6-month, TLPP at 12-months must be successful.
Time Frame: 6 months post index procedure
Population: Number of Participants with Access Circuit Primary Patency (ACPP). Modified Intended to Treat (mITT) population results were analyzed for this effectiveness endpoint. N = number of subjects in mITT population with evaluable data. Excluded subjects that discontinued, expired and or access abandoned prior to day 15.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 134 | 117
Participants | 67 | 50

5. Secondary Outcome: Number of Participants With Target Lesion Primary Patency (TLPP)
Description: Defined as the interval following the index intervention until the next clinically driven reintervention at the original treatment site or until the extremity is abandoned for permanent access.
  mITT subjects results are presented. N= number of subjects in the mITT Population with evaluable data. Evaluation through 1, 3, 18 and 24 months post index procedure.
Time Frame: 1, 3, 18 and 24 months post index procedure
Population: Number of Participants with Target Lesion Primary Patency (TLPP). Number of participants (n) in each follow-up periods varies from overall enrollment (N) as some subjects discontinued participation before the 30 days or 90 days follow-up or did not meet endpoint inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 140 | 125
Participants
  TLPP at 30-day Follow-up | 136 | 122
  TLPP at 90-day Follow-up: number analyzed (Participants) | 138 | 121
  TLPP at 90-day Follow-up | 125 | 98
  TLPP at 18 month Follow-Up: number analyzed (Participants) | 116 | 111
  TLPP at 18 month Follow-Up | 44 | 16
  TLPP at 24 month Follow-Up: number analyzed (Participants) | 114 | 110
  TLPP at 24 month Follow-Up | 40 | 10

6. Secondary Outcome: Number of Participants With Access Circuit Primary Patency (ACPP)
Description: ACPP is defined as the interval following the index intervention until the next access thrombosis or repeated intervention.
  N = number of subjects in the mITT Population with evaluable data.
Time Frame: 1, 3, 12, 18, and 24 months post index procedure
Population: Number of Participants with ACPP by Follow-up Period (mITT subjects). Number of participants (n) in each follow-up periods varies from overall enrollment (N) as some subjects discontinued participation before the 30 days and 90 days follow-up or did not meet endpoint inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 140 | 125
Participants
  ACPP at 30-day Follow-up | 133 | 120
  ACPP at 90-day Follow-up: number analyzed (Participants) | 138 | 121
  ACPP at 90-day Follow-up | 110 | 95
  ACPP at 12-month Follow-Up: number analyzed (Participants) | 128 | 114
  ACPP at 12-month Follow-Up | 33 | 19
  ACPP at 18 month Follow-Up: number analyzed (Participants) | 122 | 112
  ACPP at 18 month Follow-Up | 17 | 13
  ACPP at 24 month Follow-Up: number analyzed (Participants) | 121 | 111
  ACPP at 24 month Follow-Up | 13 | 9

7. Secondary Outcome: Number of Participants Free From Device and Procedure Related AEs Involving the AV Access Circuit
Description: Number of Participants Free from Device and Procedure Related AEs Involving the AV Access Circuit (ITT population).
  Number of participants (n) in each follow-up periods varies from overall enrollment (N) as some subjects discontinued participation before the 30 days, 90 days and 6 months follow-up or did not meet endpoint inclusion criteria.
  The relationships with device/procedure of the events are based on CEC adjudications.
Time Frame: Evaluation through 1, 3, 6, 12, 18, and 24 months post-index procedure
Population: Number of Participants Free from Device and Procedure (DP) Related AEs Involving the AV Access Circuit (ITT subjects).
  Number of participants (n) in each follow-up periods varies from overall enrollment (N) as some subjects discontinued participation before the 30 days, 90 days and 6 months follow-up or did not meet endpoint inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 140 | 137
Participants
  DP AEs Free at 30 day Follow-up | 127 | 132
  DP AEs Free at 90 day Follow-up: number analyzed (Participants) | 138 | 133
  DP AEs Free at 90 day Follow-up | 124 | 127
  DP AEs Free at 6 month Follow-up: number analyzed (Participants) | 134 | 129
  DP AEs Free at 6 month Follow-up | 118 | 122
  DP AEs Free at 12 month Follow-up: number analyzed (Participants) | 126 | 123
  DP AEs Free at 12 month Follow-up | 108 | 112
  DP AEs Free at 18 month Follow-Up: number analyzed (Participants) | 120 | 114
  DP AEs Free at 18 month Follow-Up | 99 | 102
  DP AEs Free at 24 month Follow-up: number analyzed (Participants) | 114 | 104
  DP AEs Free at 24 month Follow-up | 91 | 90

8. Secondary Outcome: Total Number of Arteriovenous (AV) Access Circuit Reinterventions
Description: Defined as the number of reinterventions to the AV access circuit until access abandonment or through study completion.
  Whereas the outcome measure time frames for the overall study are 1, 3, 6, 12,18 and 24 months, the interim report only provides the 1, 3, and 6 months results. The 12,18 and 24 months results will be provided in the final reporting for the study.
  MITT results are presented for this analysis.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: The (n) in each follow-up periods vary from overall enrollment (N) as some subjects discontinued participation before each follow-up or did not meet endpoint inclusion criteria.
  The total number of Reinterventions by Follow-Up Period was analyzed as opposed to the number of subjects with at least one AV Access Circuit Reintervention -mITT subjects
Measure: Number; unit: AV Access Circuit Reinterventions
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 112 | 107
AV Access Circuit Reinterventions
  AV Access Circuit Reinterventions at 30 days: number analyzed (Participants) | 7 | 6
  AV Access Circuit Reinterventions at 30 days | 7 | 6
  AV Access Circuit Reinterventions at 90 days: number analyzed (Participants) | 30 | 27
  AV Access Circuit Reinterventions at 90 days | 35 | 34
  AV Access Circuit Reinterventions at 6 months: number analyzed (Participants) | 69 | 71
  AV Access Circuit Reinterventions at 6 months | 103 | 107
  AV Access Circuit Reinterventions at 12 months: number analyzed (Participants) | 101 | 102
  AV Access Circuit Reinterventions at 12 months | 226 | 241
  AV Access Circuit Reinterventions at 18 months: number analyzed (Participants) | 109 | 104
  AV Access Circuit Reinterventions at 18 months | 310 | 313
  AV Access Circuit Reinterventions at 24 months | 390 | 398

9. Secondary Outcome: Total Number of Target Lesion Reinterventions
Description: Total Number of Target Lesion Reinterventions defined as the number of reinterventions to maintain target lesion patency (mITT subjects).
  Whereas the outcome measure time frames for the overall study are 1, 3, 6, 12,18 and 24 months.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: The (n) in each follow-up periods vary from overall enrollment (N) as some subjects discontinued participation before each follow-up or did not meet endpoint inclusion criteria.
  The total number of Target Lesion Reinterventions by Follow-Up Period was analyzed as opposed to the number of subjects with at least one AV Target Lesion Reintervention.
Measure: Number; unit: Target Lesion Reinterventions
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 76 | 103
Target Lesion Reinterventions
  Target Lesion Reinterventions at 30 day Follow-up: number analyzed (Participants) | 5 | 3
  Target Lesion Reinterventions at 30 day Follow-up | 5 | 3
  Target Lesion Reinterventions at 90 day Follow-up: number analyzed (Participants) | 13 | 22
  Target Lesion Reinterventions at 90 day Follow-up | 16 | 24
  Target Lesion Reinterventions 6 month Follow-up: number analyzed (Participants) | 31 | 66
  Target Lesion Reinterventions 6 month Follow-up | 40 | 92
  Target Lesion Reinterventions at 12 month Follow-Up: number analyzed (Participants) | 59 | 100
  Target Lesion Reinterventions at 12 month Follow-Up | 95 | 196
  Target Lesion Reintervention at 18 month Follow-Up: number analyzed (Participants) | 73 | 101
  Target Lesion Reintervention at 18 month Follow-Up | 139 | 248
  Target Lesion Reintervention at 24 month Follow-Up | 179 | 309

10. Secondary Outcome: Index of Patency Function (IPF)
Description: IPF is defined as the time from the index study procedure to study completion or access abandonment divided by the number of visits for a reintervention performed on the AV access circuit in order to maintain vascular access for hemodialysis. A visit is defined as one (1) procedural event, regardless of the number or type of interventions performed during the visit. The index procedure is counted as the first visit to ensure all subjects have a denominator of at least one.
  Whereas the measure time frames for the overall study are 1, 3, 6, 12,18 and 24 months.
  The IPF is representative of the number of days between interventions to maintain access circuit patency. Higher values represent a better outcome, that is, more time elapsed between the Index study procedure and reinterventions.
  mITT results are analyzed.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: Number of participants (n) in each follow-up periods varies from overall enrollment (N) as some subjects discontinued participation before the 30 days, 3 months and 6 months follow-up or did not meet endpoint inclusion criteria.
  mITT subjects results are presented.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 140 | 125
Days
  Index of Patency at 30 days Follow-up | 29.22 (3.420) | 29.28 (3.219)
  Index of Patency at 90 days Follow-up: number analyzed (Participants) | 138 | 121
  Index of Patency at 90 days Follow-up | 79.41 (20.511) | 78.98 (20.770)
  Index of Patency at 6 month Follow-up: number analyzed (Participants) | 134 | 117
  Index of Patency at 6 month Follow-up | 126.06 (54.449) | 116.11 (53.175)
  Index of Patency at 12 month Follow-up: number analyzed (Participants) | 129 | 115
  Index of Patency at 12 month Follow-up | 172.04 (108.690) | 146.09 (89.723)
  Index of Patency at 18 month Follow-up: number analyzed (Participants) | 124 | 113
  Index of Patency at 18 month Follow-up | 199.31 (145.278) | 175.70 (125.145)
  Index of Patency at 24 month Follow-up: number analyzed (Participants) | 123 | 111
  Index of Patency at 24 month Follow-up | 219.45 (178.916) | 180.59 (135.216)

11. Secondary Outcome: Index of Patency Function - Target Lesion (IPF-T)
Description: IPF-T (Index of Patency Function - Target Lesion) is defined as the time from the index study procedure to study completion or complete access abandonment divided by the number of visits for a reintervention performed at the target lesion in order to maintain vascular access for hemodialysis.
  Whereas the measure time frames for the overall study are 1, 3, 6, 12, 18 and 24 months.
  The IPF for target lesion patency is representative of the approximate (mean) number of days between interventions to maintain target lesion patency. Higher values represent a better outcome, that is, more time elapsed between the Index study procedure and reinterventions.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 140 | 125
Days
  IPTF-T at 30 days Follow-Up | 29.44 (2.958) | 29.64 (2.305)
  IPTF-T at 90 days Follow-Up: number analyzed (Participants) | 137 | 120
  IPTF-T at 90 days Follow-Up | 85.15 (15.349) | 81.35 (18.243)
  IPTF-T at 6 month Follow-Up: number analyzed (Participants) | 133 | 116
  IPTF-T at 6 month Follow-Up | 156.32 (43.724) | 121.75 (51.940)
  IPTF-T at 12 month Follow-up: number analyzed (Participants) | 122 | 114
  IPTF-T at 12 month Follow-up | 256.32 (115.626) | 160.37 (87.504)
  IPTF-T at 18 month Follow-Up: number analyzed (Participants) | 114 | 112
  IPTF-T at 18 month Follow-Up | 318.24 (179.651) | 200.64 (130.055)
  IPTF-T at 24 month Follow-Up: number analyzed (Participants) | 112 | 110
  IPTF-T at 24 month Follow-Up | 380.40 (249.548) | 217.57 (158.373)

12. Secondary Outcome: Number of Participants With Post-intervention Secondary Patency
Description: Secondary Patency is defined as the interval after the index intervention until the access is abandoned. Multiple repetitive treatments can be included in post-intervention secondary patency.
  Whereas the measure time frames for the overall study are 1, 3, 6, 12,18 and 24 months, the interim report only provides the 1, 3, and 6 months results. The 12,18 and 24 months results will be provided in the final reporting for the study.
  mITT subjects results are presented.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: Post-Intervention Secondary Patency by Follow-Up Period (mITT Subjects). (n) varies in relation to the number of failures (access abandonment) recorded at 30 days, 90 days and 6 months. Accordingly, the (n) for each period may be different from the overall (N) reported in the Participant Flow section.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 140 | 125
Participants
  Participants with Secondary Patency at 30 days | 139 | 125
  Participants with Secondary Patency at 90 days: number analyzed (Participants) | 138 | 120
  Participants with Secondary Patency at 90 days | 136 | 119
  Participants with Secondary Patency at 6 months: number analyzed (Participants) | 134 | 115
  Participants with Secondary Patency at 6 months | 131 | 113
  Participants with Secondary Patency at 12 months: number analyzed (Participants) | 122 | 105
  Participants with Secondary Patency at 12 months | 115 | 102
  Participants with Secondary Patency at 18 months: number analyzed (Participants) | 112 | 94
  Participants with Secondary Patency at 18 months | 103 | 91
  Participants with Secondary Patency at 24 months: number analyzed (Participants) | 104 | 82
  Participants with Secondary Patency at 24 months | 95 | 76

13. Secondary Outcome: Number of Participants With Technical Success
Description: Technical Success is defined as successful deployment, based on the operator's opinion, of the implant to the intended location assessed at the time of the index procedure. Therefore, for this measure, only COVERA data are relevant.
  mITT results are presented. Number of participants (n) included in this analysis is different from overall enrollment (N) as some subjects discontinued participation before the 30 days, 90 days and 6 months follow-up or did not meet endpoint inclusion criteria.
  Technical success was assessed on the day the index procedure was performed, which may be a different day for each participant.
Time Frame: On Day of Index Procedure
Population: Number of Participants with Acute Technical Success (mITT Subjects). Please note that "Technical Success is defined as successful deployment, based on the operator's opinion, of the implant to the intended location assessed at the time of the index procedure." Therefore, for this measure, only COVERA data are relevant.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera Vascular Covered Stent Following PTA
Number analyzed (Participants) | 140
Participants | 140

14. Secondary Outcome: Number of Participants With Procedure Success
Description: Procedure Success is defined as anatomic success and resolution of the pre-procedural clinical indicator(s) (clinical success) of a hemodynamically significant stenosis.
  Procedure success was assessed on the day the index procedure was performed, which may be a different day for each participant.
Time Frame: On Day of Index Procedure
Population: Procedure Success (mITT Subjects). Number of participants (n) included in this analysis is different from overall enrollment (N) as some subjects discontinued participation before the 30 days, 90 days and 6 months follow-up or did not meet endpoint inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
Number analyzed (Participants) | 140 | 126
Participants | 138 | 124

ADVERSE EVENTS:
Time Frame: Data provided for Adverse Events (AEs) and Serious Adverse Events (SAEs) at 6-Month Follow-Up Period (ITT Subjects). All subjects underwent a clinical evaluation at the index procedure: treated subjects also underwent a follow-up clinical evaluation prior to hospital discharge. Subsequent follow-up for all treated subjects was performed at 30 days, 90 days and 6 months. The 6 month follow up was an office visit to the investigational site in addition to a telephone call to dialysis centre.
Description: Both AEs and SAEs were collected based on the ITT population. SAEs results shown are CEC adjudicated.
  Note that n= subjects with at least one event. AEs and SAEs that occurred through 180 days are included. AEs and SAEs in Tables below were reported in the CSR by Organ Class only, without regards to the specific Adverse Event Terms.
Arm/Group | Covera Vascular Covered Stent Following PTA | PTA Only Using Uncoated PTA Balloon
All-Cause Mortality (participants affected / at risk) | 27/142 | 32/138
Serious Adverse Events (participants affected / at risk) | 107/142 | 110/138
Other Adverse Events (participants affected / at risk) | 119/142 | 120/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Covera Vascular Covered Stent Following PTA (N=142) | PTA Only Using Uncoated PTA Balloon (N=138)
Blood and lymphatic (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Cardiac disorders (Cardiac disorders) | 31 (31) | 40 (40)
Eye disorders (Eye disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 20 (20) | 13 (13)
General disorders and administration site conditions (General disorders) | 19 (19) | 6 (6)
Infections and Infestations (Infections and infestations) | 47 (47) | 37 (37)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 37 (37) | 34 (34)
Investigations (Investigations) | 1 (1) | 0 (0)
Metabolism and nutrition (Metabolism and nutrition disorders) | 27 (27) | 23 (23)
Muskuloskeletal and connective disorders (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6)
Nervous system (Nervous system disorders) | 14 (14) | 14 (14)
Psychiatric (Psychiatric disorders) | 1 (1) | 5 (5)
Renal and urinary (Renal and urinary disorders) | 12 (12) | 14 (14)
Respiratory, thoracic and mediastinal (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 15 (15)
Skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Vascular (Vascular disorders) | 25 (25) | 24 (24)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Covera Vascular Covered Stent Following PTA (N=142) | PTA Only Using Uncoated PTA Balloon (N=138)
Blood and lymphatic (Blood and lymphatic system disorders) | 6 (6) | 9 (9)
Cardiac (Cardiac disorders) | 39 (39) | 44 (44)
Ear and labyrinth (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Endocrine (Endocrine disorders) | 1 (1) | 3 (3)
Eye (Eye disorders) | 3 (3) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 29 (29) | 24 (24)
General disorders (General disorders) | 25 (25) | 15 (15)
Hepatobiliary (Hepatobiliary disorders) | 3 (3) | 8 (8)
Immune system (Immune system disorders) | 0 (0) | 2 (2)
Infections and Infestations (Infections and infestations) | 60 (60) | 43 (43)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 56 (56) | 45 (45)
Investigations (Investigations) | 4 (4) | 4 (4) — Electrocardiogram ST segment depression, liver function, abnormal and test abnormal, peritoneal effluent and troponin T increase.
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 33 (33) | 33 (33)
Muskuloskeletal and connective tissues (Musculoskeletal and connective tissue disorders) | 20 (20) | 12 (12)
Neoplasm benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Nervous system disorders (Nervous system disorders) | 21 (21) | 21 (21)
Psychiatric (Psychiatric disorders) | 2 (2) | 9 (9)
Renal and urinary (Renal and urinary disorders) | 13 (13) | 14 (14)
Reproductive system and breast (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 24 (24)
Skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 11 (11) | 7 (7)
Vascular (Vascular disorders) | 37 (37) | 35 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to PI publication of site results, sponsor requires publication of multi-centers results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT02649946/Prot_SAP_001.pdf